CLINICAL TRIAL: NCT06544694
Title: A Phase 3b Study to Investigate the Effect of 0.003% AR-15512 on the Ocular Surface Characteristics of Subjects With Dry Eye Disease
Brief Title: A Study to Investigate the Effect of 0.003% AR-15512 on Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEF512-E003
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye Disease
Keywords: Dry Eyes; Eye Drops
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.003% AR-15512 (Experimental): One drop in each eye twice daily for 90 days (treatment period)
  Interventions: Drug: 0.003% AR-15512
- Artificial Tears (Active Comparator): One drop in each eye twice daily for 90 days (treatment period)
  Interventions: Other: Artificial Tears

INTERVENTIONS:
Drug: 0.003% AR-15512 — Ophthalmic solution administered via topical ocular instillation
  Arms: 0.003% AR-15512
Other: Artificial Tears — Commercially available, preservative-free lubricant eye drops
  Other Names: REFRESH® Classic
  Arms: Artificial Tears

SUMMARY:
The purpose of this study is to evaluate the effect of AR-15512 ophthalmic solution 0.003% (0.003% AR-15512) on ocular surface characteristics of subjects with dry eye disease (DED).

DETAILED DESCRIPTION:
Qualified subjects will enter a 14-day run-in period, followed by a 13-week randomized treatment period, for a total individual duration of participation of approximately 15 weeks. During the run-in period, subjects will administer Artificial Tears (REFRESH® Classic) as one drop in each eye twice daily.

This is a Phase 3b study.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a previous history of DED, clinician diagnosed or patient reported, within the previous 6 months prior to the Screening visit.
* Have used artificial tears for DED symptoms within 2 months prior to the Screening visit.
* Corrected visual acuity equal to or better than logarithm Minimum angle of reflection (logMar) +0.7 (Snellen equivalent equal to or better than 20/100), as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) scale in both eyes at both the Screening and Baseline visits.
* Good general and ocular health, as determined by the investigator using medical history, ophthalmic examination and history.
* Other protocol specified inclusion criteria may apply.

Key Exclusion Criteria:

* History or presence of any ocular disorder or condition (other than DED) in either eye that would, in the opinion of the investigator, interfere with the interpretation of the study results or subject safety.
* Current evidence of other significant ophthalmic disease requiring topical medication (e.g., glaucoma, ocular hypertension), or other ophthalmic disease which the investigator believes may interfere with study findings or interpretation.
* History of ocular surgery within 1 year prior to the Screening visit; history of corneal transplant in one or both eyes.
* Use of contact lenses in either eye within 7 days prior to the Screening visit or planned use during the study.
* Regular use, as assessed by the investigator, of lid hygiene or heat masks within 14 days prior to the Screening visit or any planned use during the study.
* Use of lid heating therapy or Meibomian gland probing/therapeutic expression within 1 year prior to the Screening visit or anticipated during the study.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in goblet cell density at Day 90 | Baseline (Day 1 pre-instillation), Day 90
  Goblet cells are specialized epithelial cells that secrete mucins onto the ocular surface to help hydrate and lubricate the eye surface. Samples of conjunctiva will be collected on filter papers based on a technique called impression cytology. The filter papers will then be processed in a lab to identify the number of goblet cells. The percent change in goblet cell density at Day 90 compared to Day 1 (Baseline) will be calculated. A positive change value will indicate an improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Pharma, Study Director — Alcon Research, LLC
Locations (4):
- United States (4):
  - Butchertown Clinical Trials, Louisville, Kentucky
  - Oculus Research, Garner, North Carolina
  - Wilmington Eye, Leland, North Carolina
  - CORE, Inc., Shelby, North Carolina

IPD SHARING:
Plan to Share IPD: No